CLINICAL TRIAL: NCT05495555
Title: The Cutting Efficiency of Hybrid Tips in Different Grades of Cataract
Status: Completed | Type: Observational
Sponsor: Cataract and Laser Institute of Southern Oregon (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JS-22-001
Record Dates: First submitted 2022-08-01; First posted 2022-08-10 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- High IOP setting: Cataract removal with high IOP setting
  Interventions: Device: INTREPID® Hybrid tip
- Low IOP setting: Cataract removal with low IOP setting
  Interventions: Device: INTREPID® Hybrid tip

INTERVENTIONS:
Device: INTREPID® Hybrid tip — INTREPID® Hybrid tip for cataract removal

SUMMARY:
The objective is to assess the efficiency (as measured by phaco time, aspiration time, and fluid use) of the hybrid tip in removing cataract grade 3 & 4 in high and low intraocular pressure (IOP) settings.

DETAILED DESCRIPTION:
This study is a Single site, single-masked, randomized, prospective, observational study of the efficiency of the hybrid tip in removing cataract grade 3 & 4 in high and low intraocular pressure (IOP) settings. Subjects will be assessed pre-operatively, operatively and at 1 day and 1 week post-operatively. Clinical evaluations will include measurement of visual acuity, central corneal thickness, IOP, visual analog pain scale, and slit lamp examination.

ELIGIBILITY:
Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Be eligible to undergo sequential bilateral uncomplicated cataract surgery
* Grade 3 or 4 cataract (PNS or LOCS III)
* Undergo uneventful cataract surgery
* Gender: Males and Females.
* Age: 50 or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Patient under 50 years of age
* Unable to complete sequential bilateral cataract surgery in both eyes by the same surgeon (JS)
* Patient cataract surgery complicated by posterior capsular tear
* Any disease state deemed by PI that increases risk of complicated cataract surgery (ie Pseudoexfoliation syndrome, zonular dehiscence, history of eye trauma. RA, prior refractive surgery, etc)

The principal investigator reserves the right to declare a patient ineligible or non- evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be 50 years of age or older and who are eligible to undergo sequential bilateral uncomplicated cataract surgery.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Spaulding, DO, Principal Investigator — Cataract & Laser Institute
Locations (1):
- Cataract & Laser Institute, Medford, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | High IOP Setting | Low IOP Setting
Started | 51; 51 Eyes | 51; 51 Eyes
Completed | 51; 51 Eyes | 51; 51 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants.
Arm/Group | All Participants
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Phaco Time
Time Frame: Day 0 (surgical visit)
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | High IOP Setting | Low IOP Setting
Number analyzed (Participants) | 51 | 51
Number analyzed (Eyes) | 51 | 51
seconds | 41.6 (10) | 41.8 (10.2)

2. Primary Outcome: Aspiration Time
Time Frame: Day 0 (surgical visit)
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | High IOP Setting | Low IOP Setting
Number analyzed (Participants) | 51 | 51
Number analyzed (Eyes) | 51 | 51
seconds | 101.7 (27.2) | 106.7 (25.3)

3. Primary Outcome: Fluid Use
Time Frame: Day 0 (surgical visit)
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: Eyes
Arm/Group | High IOP Setting | Low IOP Setting
Number analyzed (Participants) | 51 | 51
Number analyzed (Eyes) | 51 | 51
mL | 41.6 (9.0) | 40.2 (7.8)

4. Secondary Outcome: Central Corneal Thickness Change From Baseline
Time Frame: baseline and 1 week postoperative
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | High IOP Setting | Low IOP Setting
Number analyzed (Participants) | 51 | 51
Number analyzed (Eyes) | 51 | 51
µm | 5.4 (5.1) | 8.1 (8.9)

5. Other Pre Specified Outcome: Cumulative Dissipated Energy
Description: This will measure the the amount of ultrasound energy used during cataract removal
Time Frame: Day 0 (surgical visit)
Measure: Mean (Standard Deviation); unit: µJ
Units Other Than Participants: Eyes
Arm/Group | High IOP Setting | Low IOP Setting
Number analyzed (Participants) | 51 | 51
Number analyzed (Eyes) | 51 | 51
µJ | 8.7 (3.1) | 8.6 (3.4)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | High IOP Setting | Low IOP Setting
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 3/51 | 3/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High IOP Setting (N=51) | Low IOP Setting (N=51)
Elevated IOP (Eye disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT05495555/Prot_SAP_000.pdf